CLINICAL TRIAL: NCT01534247
Title: A Phase I, Open-Label, 3-way Crossover, Pharmacokinetic and Drug-Drug Interaction Study of Ceftazidime Avibactam (CAZ-AVI) and Metronidazole When Administered Alone and in Combination in Healthy Subjects
Brief Title: A Study to Assess the Levels of CAZ-AVI and Metronidazole in the Blood When Given Together and Separately
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D4280C00012
Record Dates: First submitted 2012-02-09; First posted 2012-02-16 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: Phase I; drug to drug; CAZ-AVI; Healthy volunteer; pharmacokinetics; open label; metronidazole; safety
MeSH Terms: interventions — Metronidazole

ARMS (3):
- CAZAVI (Experimental): CAZ-AVI (2000 mg ceftazidime/500 mg avibactam)
  Interventions: Drug: CAZ-AVI
- Metronidazole (Active Comparator): Metronidazole (500 mg)
  Interventions: Drug: metronidazole
- CAZAVI+metronidazole (Active Comparator): CAZ-AVI (2000mg ceftazidime/500 mg avibactam) + metronidazole (500 mg)
  Interventions: Drug: CAZ-AVI + metronidazole

INTERVENTIONS:
Drug: CAZ-AVI — Infusion
  Arms: CAZAVI
Drug: metronidazole — Infusion
  Arms: Metronidazole
Drug: CAZ-AVI + metronidazole — Infusion
  Arms: CAZAVI+metronidazole

SUMMARY:
The purpose of the study is to assess whether there is any pharmacokinetic interactions between CAZ-AVI and metronidazole.

DETAILED DESCRIPTION:
A Phase I, Open-Label, 3-way Crossover, Pharmacokinetic and Drug-Drug Interaction Study of ceftazidime avibactam (CAZ-AVI) and Metronidazole when Administered Alone and in Combination in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study-specific procedures.
* Healthy male and female subjects aged 18 to 50 years (inclusive) with suitable veins for cannulation or repeated venipuncture; female subjects must be post menopausal or surgically sterile.
* Male subjects should be willing to use barrier contraception ie, condoms, from the first day of the investigational product administration until 3 months after the last administration of the investigational product.
* Have a body mass index (BMI) between 19 and 30 kg/m2
* Be able to understand and willing to comply with study procedures, restrictions, and requirements, as judged by the Investigator

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* Known history of serious allergy, hypersensitivity (eg, anaphylaxis), or any serious reaction to carbapenem or cephalosporin antibiotics or other beta-actam antibiotics or any other investigational product to be administered as part of the study
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks prior to the first administration of investigational product Any clinically significant abnormalities in physical examination, ECG, clinical chemistry, haematology, or urinalysis results, as judged by the Investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Profile of pharmacokinetic of ceftazidime, avibactam and metronidazole when administering CAZ-AVI plus metronidazole in combination compared to administration of individual components | CAZ-AVI: pre-dose, 0.5, 1, 1.5, 2, 2.25, 2.5, 2.75, 3, 4, 5, 7, 11, 23, 73, 73.5, 74, 74.5, 75, 75.25, 75.5, 75.75, 76, 77, 78, 80, 84 and 95 hours post-dose
Profile of pharmacokinetic of ceftazidime, avibactam and metronidazole when administering CAZ-AVI plus metronidazole in combination compared to administration of individual components | Metronidazole: pre-dose, 0.5, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 72, 72.5, 73, 73.25, 73.5, 74, 75, 76, 78, 80, 84 and 96 hours post-dose
Profile of pharmacokinetic of ceftazidime, avibactam and metronidazole when administering CAZ-AVI plus metronidazole in combination compared to administration of individual components | CAZ-AVI and metronidazole: pre-dose, 0.5, 1, 1.25, 1.5, 2.5, 3, 3.25, 3.5, 3.75, 4, 5, 6, 8, 12, 24, 72, 72.5, 73, 73.25, 73.5, 74, 74.5, 75, 75.25, 75.5, 75.75, 76, 77, 78, 80, 84 and 96 hours post-dose

SECONDARY OUTCOMES:
To assess safety and tolerability of CAZ-AVI and metronidazole when administered as a 2- and 1-hour infusion, respectively, every 8 hours by assessment of adverse events, lab, vital signs, ECG, physical examination | Screening up to 26 days after first dose

CONTACTS AND LOCATIONS:
Overall Officials: Mirjana Kujacic, MD, Study Chair — AstraZenecaMolndal Sweden; David Mathews, MD, Principal Investigator — QuintilesOverland Park, US; Paul Newell, Study Director — Astrazeneca Alderly UK
Locations (1):
- Research site, Overland Park, Kansas, United States

REFERENCES:
- [Background] Das S, Li J, Armstrong J, Learoyd M, Edeki T. Randomized pharmacokinetic and drug-drug interaction studies of ceftazidime, avibactam, and metronidazole in healthy subjects. Pharmacol Res Perspect. 2015 Oct;3(5):e00172. doi: 10.1002/prp2.172. Epub 2015 Aug 25. PMID 26516584
- See also: Redaction of D4280C00012 Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1458&filename=Redaction%20of%20D4280C00012%20Protocol.pdf